CLINICAL TRIAL: NCT01937091
Title: Determining the Barriers and Motivations to Clinical Trial Participation
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Janssen Services, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 13-1948; IGHID 1303
Record Dates: First submitted 2013-08-29; First posted 2013-09-09 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2014-04

CONDITIONS: HIV
Keywords: HIV; clinical trials

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Participants in trials: Participated in a trial of HAART for duration of > 48 weeks.
- Non-participants in trials: Never participated in clinical trials of HAART Must have been offered participation in a clinical trial and declined

SUMMARY:
Purpose: To comprehensively explore the barriers and motivators for participation in HIV clinical trials in a purposive sample of HIV positive patients receiving care at the UNC ID (Infectious Diseases) clinic Participants: HIV positive patients seen at the UNC ID Clinic. Participants will be purposively sampled based on gender, race and previous participation in HIV clinical trials. Blacks and patients who have never participated in clinical trials will be oversampled.

Procedures (methods): Cross-sectional study using in-depth semi-structured qualitative interviews to determine the barriers and motivators for participation in HIV clinical trials. Patient interviews will be audiotaped, transcribed verbatim and analyzed using Atlas.ti software to understand the barriers and motivators for participation in HIV clinical trials.

DETAILED DESCRIPTION:
Study Population: 48 HIV positive adult (at least 18 years of age) patients receiving care at the UNC ID Clinic will be enrolled in the study. Purposive sampling by race, gender and previous participation in HIV clinical trials will be used to ensure adequate representation in each category. Participation in a clinical trial will be defined as having participated in a trial of highly active antiretroviral therapy (HAART) for duration of > 48 weeks. Non-trial participation will be defined as having been offered the opportunity to participate in a clinical trial but have never participated in any clinical trial or participated in a trial that included a one-time sample collection with no follow up visits.

STUDY METHODS

Questionnaire: The questionnaire consists of open-ended questions to be administered to participants. The questionnaire items were composed by reviewing related studies. Two versions of the questionnaire will be administered, one for participants with a history of participation in clinical trials and one for participants who were approached but have never been in a clinical trial (See Appendix 1.) The questionnaire will be revised after pre-testing to incorporate changes before it will be administered to all 48 participants.

Interview: The interview will be conducted at the UNC ID clinic by one research assistant. The interview will take approximately 45 minutes and will be audiotaped.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive adults,
* at least 18 years of age,
* receiving care at the UNC ID clinic,
* have previously been approached for (or offered) participation in a clinical trial.

Exclusion Criteria:

* Non native English speaking patients
* Unable to provide informed consent
* Have never been offered participation in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-positive adults, > 18 years, who receive care at the UNC ID clinic and who have previously been approached for (or offered) participation in a clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Reasons why people choose to or not to participate in HIV Clinical Trials based on questionnaire responses | Administered immediately following provision of informed consent

CONTACTS AND LOCATIONS:
Overall Officials: Prema Menezes, Ph. D, PA-C, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States